CLINICAL TRIAL: NCT07191431
Title: A Clinical Study on the Efficacy and Safety of Methotrexate (MTX) or Thiotepa (for MTX Intolerance) or Temozolomide (TMZ) Combined With Orelabrutinib and Selinexor in Relapsed/Refractory Primary or Secondary Central Nervous System Lymphoma（SELINA）
Acronym: SELINA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SELINA
Record Dates: First submitted 2025-09-04; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Lymphoma Cns
Keywords: lymphoma CNS; Selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- selinexor (Experimental): inductive treatment
  * Orelabrutinib 150mg qd + Selinexor 40mg qw
  * Combined chemotherapy (choose one):
    * MTX 3.5g/m² IV d0
    * Temozolomide 150mg/m² PO d1-5
    * Thiotepa 40mg/m² IV d3
  * Every 3 weeks for 6 cycles maintenance treatment
  * Non-transplant patients: Orelabrutinib ± Selinexor (based on TP53 mutation status)
  Interventions: Drug: Selinexor+Orelabrutinib+Methotrexate/Thiotepa/Temozolomide

INTERVENTIONS:
Drug: Selinexor+Orelabrutinib+Methotrexate/Thiotepa/Temozolomide — * Orelabrutinib 150mg qd + Selinexor 40mg qw
  * Combined chemotherapy (choose one):
    * MTX 3.5g/m² IV d0
    * Temozolomide 150mg/m² PO d1-5
    * Thiotepa 40mg/m² IV d3
  * Every 3 weeks for 6 cycles

SUMMARY:
Clinical Study on the Efficacy and Safety of Methotrexate (MTX) or Thiotepa (for MTX intolerance) or Temozolomide (TMZ) Combined with Orelabrutinib and Selinexor in the Treatment of Relapsed/Refractory Primary or Secondary Central Nervous System Lymphoma

This study adopts an open-label, prospective, single-arm, single-center design aimed at evaluating the efficacy and safety of methotrexate (MTX) or thiotepa (for MTX intolerance) or temozolomide (TMZ) combined with orelabrutinib and selinexor in the treatment of relapsed/refractory primary or secondary central nervous system lymphoma (r/r CNSL).

Primary Objective To evaluate the efficacy and safety of methotrexate (MTX) or thiotepa (for MTX intolerance) or temozolomide (TMZ) combined with orelabrutinib and selinexor in the treatment of relapsed/refractory primary or secondary central nervous system lymphoma (r/r CNSL).

Secondary Objective To assess the benefit-risk balance of methotrexate (MTX) or thiotepa (for MTX intolerance) or temozolomide (TMZ) combined with orelabrutinib and selinexor in combination with chemotherapy in the clinical management of relapsed/refractory primary or secondary central nervous system lymphoma (r/r CNSL).

Patients with relapsed/refractory primary or secondary CNSL (PCNSL/SCNSL) who meet the inclusion criteria will be enrolled. Previous study data indicate that the combination of orelabrutinib with methotrexate or temozolomide in the treatment of relapsed/refractory central nervous system lymphoma can achieve an ORR of 60%. It is anticipated that the addition of selinexor will increase the ORR to 75%. The treatment effect in r/r CNSL patients is expected to be superior to that of chemotherapy-based combination regimens (one-sided test). With a one-sided alpha = 0.025, beta = 0.1, and an expected enrollment completion within 12 months, along with a follow-up period of 24 months, the planned sample size is 23 patients. Accounting for a 10% dropout rate, the corrected sample size for this study is 25 patients.

Patients who meet the inclusion/exclusion criteria and provide signed informed consent will be enrolled in the experimental group. Each treatment cycle lasts 3 weeks. After 6 cycles of induction therapy, patients who do not achieve a PR or experience disease progression at any time will withdraw from the study and receive salvage therapy. Patients who achieve CR or PR will undergo autologous transplantation if they are young and eligible for transplantation. For patients with TP53 mutations, selinexor will be incorporated into the transplant conditioning regimen. Patients who are ineligible for transplantation will receive consolidative radiotherapy. After consolidative therapy, maintenance treatment with orelabrutinib may be administered based on treatment response and patient tolerance. For patients with TP53 mutations, selinexor will be added to orelabrutinib maintenance therapy. For patients with SD/PD, subsequent treatment will be determined by the investigator, followed by observation and follow-up for up to 3 years.

Experimental Group Regimen:

Induction Therapy: Orelabrutinib 150 mg once daily, selinexor 40 mg weekly, methotrexate 3.5 g/m² (for patients intolerant or resistant to methotrexate: temozolomide 150 mg/m² or thiotepa 30-40 mg/m² may be used as alternatives). Each cycle lasts 3 weeks, for a total of 6 cycles.

Maintenance Therapy:

Non-TP53mut patients without transplantation: After consolidative radiotherapy, maintenance therapy with orelabrutinib 150 mg once daily may be administered.

TP53mut patients without transplantation: After consolidative radiotherapy, maintenance therapy with orelabrutinib 150 mg once daily combined with selinexor 40 mg weekly may be administered.

DETAILED DESCRIPTION:
1. Research Background

   1.1 Significance of the Research Central nervous system lymphoma (CNSL) is a rare extranodal non-Hodgkin lymphoma characterized by high aggressiveness and poor prognosis. Over the past decades, high-dose methotrexate (HD-MTX)-based chemotherapy regimens (including combinations with rituximab, temozolomide, cytarabine, vincristine, etc.) have significantly improved the survival outcomes of CNSL patients . However, treatment options for relapsed/refractory primary and secondary central nervous system lymphoma (r/r CNSL) remain limited, necessitating the exploration of new combination therapies. This project aims to conduct a single-center, randomized, open-label, single-arm clinical trial of orelabrutinib combined with chemotherapy for r/r CNSL, analyzing patients' short- and long-term efficacy and chemotherapy-related toxic side effects, ultimately providing a reference for further optimizing the treatment of r/r CNSL.

   1.2 Research Background Central nervous system lymphoma includes primary central nervous system lymphoma (PCNSL) and secondary central nervous system lymphoma (SCNSL). PCNSL is a relatively rare type of non-Hodgkin lymphoma (NHL) originating in the central nervous system (including the brain, eyes, spinal cord, and meninges) without involvement of other sites. It accounts for about 2%-4% of all intracranial tumors and 4%-6% of all NHLs, and its incidence has been gradually increasing in recent years . SCNSL refers to lymphoma that spreads to the CNS during or after treatment for systemic lymphoma. It can be diagnosed at the initial diagnosis of lymphoma or at relapse .

   Over the past decades, HD-MTX-based chemotherapy regimens (including rituximab, temozolomide, cytarabine, vincristine, etc.) have significantly improved the survival prognosis of PCNSL patients, but the relapse rate exceeds 50%, and about 25% of patients fail initial treatment. The prognosis for r/r PCNSL is even worse . Furthermore, retrospective studies show that the median survival of previously treated SCNSL patients is approximately 6 months .

   Due to the poor survival of patients, prospective studies for r/r CNSL patients are lacking; current knowledge is based on retrospective studies of cytotoxic drugs or combination regimens used to treat systemic lymphoma . In one retrospective study, 22 r/r CNSL patients who had initially received high-dose methotrexate-based chemotherapy were treated with a combination of rituximab, ifosfamide, and etoposide for 4 cycles. The ORR was 41%, CR rate was 37%, and the 2-year PFS was 21% .

   Temozolomide is a well-tolerated oral alkylating agent that has shown activity in other brain tumors, with CNS concentrations about 20% lower than corresponding blood concentrations . A prospective study showed that temozolomide monotherapy for r/r CNSL patients achieved an ORR of only 31% .

   It is known that in CNSL tumor cells, the B-cell receptor pathway and MYD88 gene often mutate, leading to sustained activation of the nuclear factor-kappa B (NF-κB) signaling pathway . Bruton's tyrosine kinase (BTK) is a key regulatory molecule in the B-cell receptor pathway and is considered one of the ideal targets for treating lymphoma with sustained NF-κB pathway activation . For CNSL, a preclinical study reported that ibrutinib achieves high drug levels in the brain, suggesting that the BTK inhibitor ibrutinib might be effective against central lymphoma . Subsequently, two clinical trials found that the objective response rate (ORR) in relapsed PCNSL patients receiving ibrutinib combined with chemotherapy could reach 75% . These results suggest that BTK inhibitors combined with existing chemotherapy regimens may help improve patient ORR and ultimately enhance the survival prognosis of these patients. However, due to ibrutinib's off-target effects which cause relatively high toxicity events, applying a new-generation BTK inhibitor with longer efficacy and lower toxicity is significant and may be more suitable for combination therapy in r/r CNSL patients.

   Orelabrutinib is a second-generation BTK inhibitor. Due to its excellent efficacy and low toxicity, it has been approved for adult patients with mantle cell lymphoma (MCL) who have received at least one prior therapy; adult patients with chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL) who have received at least one prior therapy; and relapsed/refractory marginal zone lymphoma (MZL) . A phase II clinical study found that in r/r PCNSL patients, the median cerebrospinal fluid (CSF) concentration of orelabrutinib was 28.7 ng/ml (range, 11.8-52.7 ng/ml), with a median CSF/plasma free ratio of 59.8% (range 46.09%-86.67%). This result indicates that orelabrutinib can effectively cross the blood-brain barrier (BBB) . Furthermore, Yang C et al. reported that an orelabrutinib combination regimen (orelabrutinib + lenalidomide + RMT) achieved an ORR of 86.7% in 15 r/r PCNSL patients, with a median PFS of 9.8 months . Thus, orelabrutinib has potential application prospects in the treatment of r/r CNSL, and the efficacy and safety of orelabrutinib combination regimens for treating r/r CNSL warrant further exploration.

   Selinexor is a Selective Inhibitor of Nuclear Export (SINE), belonging to a new class of targeted anticancer drugs. Its mechanism of action involves specifically inhibiting Exportin 1 (XPO1), blocking the transport of tumor suppressor proteins, growth regulators, and anti-inflammatory proteins from the nucleus to the cytoplasm. This causes the accumulation of these key proteins within the nucleus, thereby inducing cancer cell apoptosis and inhibiting tumor growth.

   Therefore, this study plans to conduct a single-center, randomized, open-label, single-arm clinical trial of methotrexate (MTX) or thiotepa (for MTX intolerance) or temozolomide (TMZ) combined with orelabrutinib and selinexor for the treatment of r/r CNSL, analyzing patients' short- and long-term efficacy and chemotherapy-related toxic side effects, ultimately providing a reference for further optimizing the treatment of r/r CNSL.
2. Study Design

2.1 Overall Design This study adopts an open-label, prospective, single-arm, single-center design aimed at evaluating the efficacy and safety of orelabrutinib combined with chemotherapy in r/r CNSL.

2.2 Definition of Study Endpoints

Primary Endpoint Objective Response Rate (ORR)

Secondary Endpoints 2-year Progression-Free Survival (PFS) rate; Overall Survival (OS); Complete Response (CR) rate; Safety.

Safety endpoints: Incidence and grade of adverse events (AEs) and serious adverse events (SAEs); ECOG performance status, vital signs, physical examination, laboratory test indicators, electrocardiogram (ECG), echocardiogram, etc.; Incidence of thrombotic events.

Exploratory Endpoints Blood and cerebrospinal fluid concentrations of selinexor;

Cerebrospinal fluid and peripheral blood ctDNA:

Collect patient cerebrospinal fluid (4ml each time) at four time points: pre-treatment, before cycle 2, end of treatment, and at disease progression.

Peripheral blood anticoagulant sample (4ml), once during follow-up; Extract circulating tumor DNA (ctDNA), using capture and next-generation sequencing technology, Capp-seq for detection, analyzing the correlation of ctDNA with tumor burden, molecular mutations, molecular response, and for prognosis, treatment response, relapse, and drug resistance. Single-cell sequencing will be performed on some patients for deeper research.

2.3 Determination of Sample Size

Based on historical data showing an ORR of approximately 41% for chemotherapy combination regimens in r/r CNSL patients, combined with research and current clinical needs, where ibrutinib combined with chemotherapy showed 69% efficacy in r/r CNSL, and considering orelabrutinib's higher concentration across the blood-brain barrier and potentially better effect, it is hypothesized that this study's ORR will increase to 75%. The treatment effect in r/r CNSL patients is expected to be superior to that of chemotherapy combination regimens (one-sided test). With a one-sided alpha = 0.025, beta = 0.1, an expected enrollment completion within 12 months, and a follow-up period of 24 months, the planned sample size is 23 patients. Accounting for a 10% dropout rate, the corrected sample size for this study is 25 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria to be enrolled in this study:
* Fully understand this study and voluntarily sign the informed consent form;
* Age: 14-80 years;
* Life expectancy judged by the investigator to exceed 3 months;
* B-cell origin central nervous system lymphoma (CNSL) confirmed by pathology or flow cytometry (histology or cytology);
* Relapsed or refractory PCNSL or SCNSL: Must have received at least one prior systemic therapy for CNS lesions; number of relapses is not restricted;
* Any non-hematological toxicity related to prior treatment should have recovered to Grade 1 or normal (according to NCI CTCAE version 5.0, except alopecia).
* Bone marrow and organ function meeting the following criteria (no transfusion, no G-CSF use, no medication for correction within 14 days before screening):

Bone marrow function: Absolute neutrophil count ≥1.0x10⁹/L, platelets ≥50x10⁹/L, hemoglobin ≥60g/L;Liver function: Serum total bilirubin ≤1.5xULN (≤3.0xULN if liver metastases present); AST and ALT ≤ 2.5xULN (≤5.0xULN if liver metastases present);Coagulation function: International Normalized Ratio (INR) and activated partial thromboplastin time ≤1.5xULN;Renal function: Serum creatinine ≤1.5xULN or estimated creatinine clearance ≥30 mL/min (Male: Cr (mL/min) = (140 - age) x weight (kg) / (72 x serum creatinine (mg/dL)); Female: Cr (mL/min) = (140 - age) x weight (kg) / (85 x serum creatinine (mg/dL))).

* Female subjects of childbearing potential and male subjects with reproductive ability, who have no pregnancy plan with their partners during the study period and for 3 months after treatment interruption, must use one of the following effective contraceptive methods throughout the study and for 3 months after treatment interruption: abstinence, physical contraception (e.g., ligation, condoms, etc.), hormonal contraceptive drugs started at least 3 months before the first dose in the study. Male subjects are prohibited from sperm donation from the start of treatment until 3 months after treatment cessation. The patient or their legal guardian voluntarily signs the informed consent form.
* Good compliance, willing to adhere to the visit schedule, dosing plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

* Patients who meet any of the following criteria will not be allowed to enter this study:
* Contraindication to any drug in the treatment regimen;
* Subject has a history of active liver disease, including viral or other hepatitis or cirrhosis (Hepatitis B defined as HBV-DNA above the upper limit of normal; active Hepatitis C defined as seropositive for HCV antibody, but those with negative HCV-RNA can be enrolled);
* Human Immunodeficiency Virus (HIV) infection;
* Congestive heart failure (New York Heart Association Class >2); history of acute myocardial infarction, unstable angina, stroke, or transient ischemic attack within the past six months;
* Hereditary long QT syndrome or QTc >480ms (Note: QTc interval must be calculated using Fridericia's formula, QTcF = QT/(RR)^0.33);
* Pregnant and lactating women, or those planning to become pregnant during the study period;
* Clear history of neurological or psychiatric disorders, or history of psychotropic drug abuse or drug addiction;
* Clinically significant active infection.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2027-09-02 (Estimated); Study Completion 2029-09-02 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 6 months
  Optimal response rates during the treatment period

SECONDARY OUTCOMES:
2-year Progression-Free Survival Rate | up to 2 years
  the probability of no tumor progression (such as tumor enlargement or new lesions) within 2 years after treatment.

OTHER OUTCOMES:
CRR | up to 6 months
  Number of subjects who achieve complete remission during treatment
OS | up to 3 years
  Refers to the time from the start of randomization to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes